CLINICAL TRIAL: NCT00128297
Title: Randomized, Multicentric Phase IV Clinical Trial for the Administration of Pamidronate in Breast Cancer Patients With Bone Metastases
Brief Title: Pamidronate Administration in Breast Cancer Patients With Bone Metastases
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Spanish Breast Cancer Research Group (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GEICAM 2000-01
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Neoplasm Metastasis
Keywords: Breast cancer patients with symptomatic bone metastases
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis | interventions — Pamidronate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A: continuous administration (Active Comparator): Pamidronate 90 mg/m2 iv every 3-4 weeks, during 18 months
  Interventions: Drug: Pamidronate
- Arm B: alternate administration (Experimental): Pamidronate 90 mg/m2 iv every 3-4 weeks, during 6 months, followed by a 6 month rest, and a new 6 months treatment period.
  Interventions: Drug: Pamidronate

INTERVENTIONS:
Drug: Pamidronate
  Other Names: Aredia

SUMMARY:
The study objective is to evaluate the differences, in terms of first occurrence of a skeletal event, in patients with breast cancer and symptomatic bone metastases, when pamidronate is administered during 2 years, or when it is administered during 6 months, followed by a six month rest period, and again a 6 month treatment period.

DETAILED DESCRIPTION:
Background: Pamidronate (PMT) is effective in reducing skeletal related events (SRE) in breast cancer (BC) patients with bone metastasis (BM). Its best way of administration and optimum treatment duration are still to be determined.

Objective: evaluate the efficacy of continuous administration (arm A) vs. alternate administration (arm B) of PMT to delay time to first SRE in BC pt presenting with symptomatic BM.

Methods: patients aged >18, Eastern Cooperative Oncology Group (ECOG) performance status ≥ 2, adequate renal function, and BC symptomatic BM were eligible. BM was defined as presence of 3 or more hot spots (HS) in skeletal scintigraphy (SS), or any number of HS in SS if osteolytic, osteoblastic or mixed bone lesions determined by radiography, or 2 or less HS in SS if magnetic resonance or CT scan confirmation of BM. Symptomatic BM was defined as pain associated to SS HS, or SRE (pathological fractures or spine cord compression or radiation bone treatment or tumour induced hypercalcemia), or treatment with analgesia due to bone pain. Patients were allowed up to 1 previous chemotherapy and 2 previous hormone therapy lines for metastatic disease. Antineoplastic therapy could be changed at any time during the study. Eligible patients were stratified (isolated bone metastasis or associated to node or skin lesions vs. bone metastasis associated to visceral disease) and randomized to receive 2 hour-iv. PMT 90 mg every 3-4 weeks for 18 months (arm A) or iv. PMT 90 mg every 3-4 weeks for 6 months, followed by a 6 months rest, and a new 6 months on-treatment period (arm B). Quality of Life (QoL) was measured with short form (SF)-36 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Up to two previous or current hormone therapy treatments for metastatic breast cancer are allowed.
* Normal or borderline renal function (serum creatinine < 1.5 x upper normal limit [UNL]).
* Normal calcium levels in serum, or slightly non-symptomatic high levels (< 1.25 x UNL).
* Performance status 0, I or II in World Health Organization (WHO) scale.

Exclusion Criteria:

* Treatment with bisphosphonates in the 30 previous days, or any time if the indication was treatment of metastatic bone lesions.
* Treatment with bisphosphonates is only allowed if the indication is hypercalcaemia.
* Metastases in central nervous system (CNS).
* Hypersensitivity to bisphosphonates or other components of the formula.
* Pregnant or lactating women.
* Previous or current treatment with a second chemotherapy line or a third hormone therapy line for metastatic disease.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2000-10-18 (Actual); Primary Completion 2004-06-04 (Actual); Study Completion 2004-06-04 (Actual)

PRIMARY OUTCOMES:
Pamidronate efficacy to prevent first skeletal event: time until the appearance of the first skeletal event | 18 months
  The main variable of evaluation is the time until the appearance of the first skeletal event. Skeletal event is defined as pathological bone fracture, or spine cord compression, or radiation bone treatment, or tumour induced hypercalcemia

SECONDARY OUTCOMES:
Number of skeletal events per treatment arm | 18 months
  The main variable of evaluation is the time until the appearance of the first skeletal event per arm.
Quality of life: Short Form (SF)-36 questionnaire | 18 months
  Quality of Life (QoL) was measured with Short Form (SF)-36 questionnaire, which is a 36 item, patient-reported survey of patient health. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score, the more disability, and the higher the score the less disability (a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability). The eight sections are vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. It will be completed since baseline visit and during all treatment period delivered to the patient before the start of each visit.
Overall survival (OS) | 18 months
  OS will be determined from the date of randomization until the date of death for any reason.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau; Study Director, Study Director — Hospital Clínico Universitario de Valencia
Locations (1):
- Spanish Breast Cancer Research Group (GEICAM), San Sebastián de los Reyes, Madrid, Spain

REFERENCES:
- See also: "Click here for more information about this study:" — http://www.geicam.org